CLINICAL TRIAL: NCT06003361
Title: Randomized Controlled Trial of a Digital Cognitive Behavioral Therapy Program for Major Depression in Adults
Brief Title: Rise Study for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Big Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-D-02
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Digital CBT (Experimental): digitally-delivered CBT for depression accessed via mobile app
  Interventions: Device: Digital CBT
- Waitlist (Other): Participants will wait for 5 weeks prior to receiving the intervention
  Interventions: Other: Waitlist

INTERVENTIONS:
Device: Digital CBT — An app-based intervention based on principles from cognitive behavioral therapy for depression.
  Arms: Digital CBT
Other: Waitlist — Participants will wait for 5 weeks prior to receiving the intervention
  Arms: Waitlist

SUMMARY:
This study will examine the efficacy of digital CBT versus waitlist in improving symptoms for adults with Major Depressive Disorder.

DETAILED DESCRIPTION:
This study aims to examine the effectiveness of app-based digital CBT in individuals with a diagnosis of Major Depressive Disorder. The primary outcomes are depression symptom reduction and engagement with fulfilling activities after 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥22 years old
* Score ≥10 and <20 on the 8-item Patient Health Questionnaire (PHQ-8)
* Diagnosis of Major Depression
* Current resident of the USA
* Oral and written fluency in English
* Regular access to the internet via a mobile or tablet device using Android (5 or higher) or iOS (13 or higher)
* Participant is able and willing to comply with protocol requirements, has been informed of the nature of the study, and has signed the IRB-approved informed consent form

Exclusion Criteria:

* Must not be currently receiving or be expecting to start therapy for depression, anxiety, or sleep during study participation, or have received cognitive behavioral therapy for depression, anxiety, or sleep in the past 12-months
* If on psychotropic medication, this must be stable for at least 60 days
* Past or present psychosis, schizophrenia, or bipolar disorder
* Moderate or greater suicide risk
* Treatment-resistant depression
* Hearing or vision impairment that prevents effective use of the audio-visual content of digital CBT or psychoeducation
* Intellectual disability or any Neurocognitive or Neurodevelopmental disorder that would prevent participants from following study procedures
* Any condition that the investigator believes would make participation in the study not in the best interest of the subject or would preclude successful completion of study activities
* Other exclusion criteria may apply

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | 5 weeks post-randomization
  Validated questionnaire; an 8-item scale with total scores between 0 and 24 where higher scores indicate greater severity
Environmental Reward Observation Scale (EROS) | 5 weeks post-randomization
  A validated 10 item scale with total scores between 10 and 40 where higher scores indicate greater engagement with rewarding or fulfilling life activities

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | 10 weeks post-randomization
  Validated questionnaire; an 8-item scale with total scores between 0 and 24 where higher scores indicate greater severity
Montgomery-Åsberg Depression Rating Scale (MADRS) | 5 and 10 weeks post-randomization
  A validated 10 item observer-rated scale with total scores between 0 and 60 where higher scores indicate greater severity
World Health Organization 5-item Wellbeing Index (WHO-5) | Weeks 5 and 10 post-randomization
  Validated questionnaire; a 5-item scale with raw total scores between 0 and 25 where higher scores indicate greater wellbeing
Environmental Reward Observation Scale (EROS) | 10 weeks post-randomization
  A validated 10 item scale with total scores between 10 and 40 where higher scores indicate greater engagement with rewarding or fulfilling life activities

CONTACTS AND LOCATIONS:
Locations (1):
- Big Health Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No